CLINICAL TRIAL: NCT06418451
Title: To Compare the Clinical Efficacy and Complications of Modified Ischial Spinous Fascia Fixation and Sacrospinous Ligament Fixation in the Treatment of Pelvic Organ Prolapse
Brief Title: A Randomized Controlled Trial of Modified Ischial Spinous Fascia Fixation and Sacrospinous Ligament Fixation in the Treatment of Pelvic Organ Prolapse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lan Zhu (Other)
Responsible Party: Sponsor-Investigator, Lan Zhu, Director of the Department of Obstetrics and Gynecology at Peking Union Medical College Hospital, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K5788
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacrospinous ligament fixation (SLFF) (Active Comparator)
  Interventions: Procedure: sacrospinous ligament fixation (SLFF)
- modified ischial spinous fascia fixation (modified ISFF) (Experimental)
  Interventions: Procedure: modified ischial spinous fascia fixation (modified ISFF)

INTERVENTIONS:
Procedure: sacrospinous ligament fixation (SLFF) — SSLF is a surgical procedure used to treat vaginal apex prolapse by fixing the vaginal apex to the right sacrospinous ligament. The procedure involves marking and incising the posterior vaginal wall, dissecting the vaginal rectal space, and placing sutures on the outer one-third of the ligament. These sutures connect the vaginal apex to the attachment point of the right uterosacral ligament. Anterior/posterior vaginal wall repair procedures can be performed if needed, without using implant materials. SSLF provides enhanced support for the vaginal apex.
  Arms: sacrospinous ligament fixation (SLFF)
Procedure: modified ischial spinous fascia fixation (modified ISFF) — The modified ISFF procedure involves making a midline incision along the posterior fornix of the vagina, exposing the ischial spine fascia. Two sutures are placed around the ischial spine and passed through the mucosa of the anterior and posterior vaginal walls, lifting the vaginal apex and anterior wall towards the spine. The procedure also allows for additional anterior/posterior vaginal wall repair if necessary, without using implant materials.
  Arms: modified ischial spinous fascia fixation (modified ISFF)

SUMMARY:
Background: Pelvic organ prolapse is one of the most common benign gynecological disorders in middle-aged and elderly women, and it has a significant negative impact on women's social, physical, and psychological health. Sacrospinous ligament fixation (SSLF) is one of the main surgical procedures for reconstructing pelvic floor defects. In previous studies, the ischial spine fascia fixation (ISFF) technique developed by our team has been shown to be a safe and effective alternative to SSLF. However, both procedures have inadequate support for the anterior vaginal wall. Therefore, based on the traditional ISFF, we fix the anterior vaginal wall to the ipsilateral ischial spine fascia to enhance support for the anterior vaginal wall. This modified procedure is called modified ISFF. This trial aims to compare the subjective and objective therapeutic effects, recurrence rates, quality of life, perioperative parameters, and complications of modified ISFF and SSLF in the treatment of patients with pelvic organ prolapse of degrees II-IV.

Methods: This trial is a randomized controlled multicenter non-inferiority trial. The primary outcome measure is the composite surgical success rate at one-year follow-up, defined as the absence of subjective vaginal bulge symptoms, no need for retreatment, and absence of POP-Q points at or beyond the hymen or vaginal introitus, i.e., Aa, Ba, C, Ap, Bp all < 0 cm. The secondary outcomes include anatomical outcomes of each vaginal segment based on the POP-Q score, subjective improvement in quality of life evaluated by questionnaires (PFIQ-7, PFDI-20, PISQ-12, and PGI-I), perioperative parameters (operation time, blood loss, length of hospital stay, pain VAS score, hospital costs), and complications. Data analysis will be conducted according to the intention-to-treat principle. Based on a composite success rate of 88% and a non-inferiority margin of -10% (one-sided α = 0.025, β = 0.2), 370 patients will be recruited from 9 centers, including a 10% dropout rate. The purpose of this study is to investigate whether modified ISFF is non-inferior to SSLF in terms of clinical efficacy and complications.

Discussion: This multicenter non-inferiority trial will evaluate the effectiveness and safety of modified ISFF compared to SSLF in symptomatic patients with degrees II-IV uterovaginal prolapse. If modified ISFF is proven to be non-inferior to SSLF, it would be a preferable alternative for patients with a shorter vaginal length and those who have difficulties with SSLF due to anatomical factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic mid-pelvic organ prolapse (POP-Q stage ≥ II) who may concurrently have anterior and/or posterior pelvic organ prolapse.
* Patients willing to undergo long-term follow-up for at least one year.
* Patients willing to sign an informed consent form and participate in this study.

Exclusion Criteria:

* Patients who have undergone previous POP or urinary incontinence surgery with the use of implant materials.
* Patients who require simultaneous anti-urinary incontinence surgery for the current procedure.
* Contraindications for general anesthesia and surgical intervention, such as severe medical comorbidities that render the patient unable to tolerate surgery.
* Patients who wish to preserve the uterus.
* Patients in the active phase of genital, urinary, or systemic infections.
* Patients who, for other reasons (such as having genital malignancies), choose not to undergo SSLF/modified ISFF surgical intervention at the moment.
* Patients who are unable or unwilling to attend follow-up visits (excluding those who may be willing to participate in telephone follow-up).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The composite success rate | At the one-year follow-up
  1. No sensation of vaginal bulge or protrusion, indicated by a response of "no" or a score of 0 on question 3 of the PFDI-20 questionnaire, which asks, "Do you often see or feel a bulge or something falling out of your vagina?"
  2. No further treatment (surgical or non-surgical) required for POP (Pelvic Organ Prolapse).
  3. Absence of POP-Q points at the hymen or beyond the hymen, indicating that Aa, Ba, C, Ap, and Bp are all < 0cm.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No